CLINICAL TRIAL: NCT05123365
Title: An Optimal Dose Finding Study of N-Acetylcysteine in Patients with Myeloproliferative Neoplasms
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Angela G. Fleischman, Associate Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20216930; UCI 20-50 (Other: CFCCC)
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Myeloproliferative Neoplasm; MPN; Essential Thrombocythemia; Polycythemia Vera; Myelofibrosis
Keywords: MPN; Myeloproliferative Neoplasm; Essential Thrombocytemia; Polycythemia Vera; Myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 1 (DL1) (Experimental): Patients take N-Acetylcysteince 600 mg orally twice daily.
  This is the starting dose level for the study.
  Interventions: Drug: N-Acetylcysteine
- Dose Level 2 (DL2) (Experimental): Patients take N-Acetylcysteince 1200 mg orally twice daily.
  If DL1 is well tolerated, the next cohort will progress to this dose level.
  Interventions: Drug: N-Acetylcysteine
- Dose Level 3 (DL3) (Experimental): Patients take N-Acetylcysteince 1800 mg orally twice daily.
  If DL2 is well tolerated, the next cohort will progress to this dose level.
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — Given PO
  Other Names: N-AC

SUMMARY:
This is a phase I/II study evaluating the optimal dose of N-acetylcysteine (N-AC) in patients with myeloproliferative neoplasms (MPN).

DETAILED DESCRIPTION:
This is a phase I/II open-label clinical trial determining the optimal biological dose (OBD) of N-acetylcysteine in subjects with myeloproliferative neoplasms. These are subjects who have a diagnosis of essential thrombocythemia (ET), polycythemia vera (PV), or myelofibrosis (MF).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Have a diagnosis of essential thrombocythemia (ET), polycythemia vera (PV), or myelofibrosis (MF) according to the 2016 WHO criteria
* Has not taken interferon-alpha or a JAK inhibitor (such as ruxolitinib or fedratinib) for treatment of MPN in the past 28 days before enrollment.
* May continue on current MPN treatment, including aspirin, hydroxyurea, or anagrelide. Therapeutic phlebotomies should continue per the patient's usual regimen.
* Has not taken N-Acetylcysteine (N-AC) or preparations containing N-AC in the past 28 days before enrollment.
* Baseline MPN-TSS score of ≥ 10 at the time of enrollment.
* Peripheral blast count <10% during Screening.
* Free of other active or metastatic malignancies other than localized skin cancer.
* Amenable to blood draws and symptom assessments.
* Agree to the use of contraceptives. Female subjects of childbearing potential and their male partners, or male subjects who have female partners of childbearing potential, should both use an effective contraception method during the study and continue to use contraception for 60 days after the last dose of study drug.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) questionnaire score of ≥3
* Currently pregnant or planning on being pregnant within the study period.
* Currently breastfeeding.
* Known uncontrolled active viral or bacterial infection.
* Significant impairment of major organ function defined as

  1. Serum creatinine clearance less than 50 ml/min (calculated with Cockroft-Gault formula).
  2. Bilirubin more than 1.5 mg/dl except for Gilbert's disease. ALT or AST more than 2X upper normal limit or has radiologic evidence of liver cirrhosis.
  3. Platelets < 100 × 10^9/L
  4. Hgb < 10 g/dL
  5. ANC < 0.75 × 10^9/L
* Known history of allergic reaction to N-AC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Optimal Biological Dose (OBD) of N-Acetylcysteine | From the start date of treatment until 7 days after completion of treatment or removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, up to 8 weeks.
  Determination of the optimal biological dose (OBD) will be utilized to evaluate the safety and tolerability of N-AC as a treatment for patients with MPN. Optimal biological dose is defined as the therapeutic dose that possesses the highest efficacy probability while inducing acceptable toxicity
Proportion of subjects who achieve 30% reduction of MPN-SAF Total symptom score (MPN-TSS) | 7 days prior to beginning treatment until end of treatment, average of 9 weeks.
  MPN-SAF Total symptom score (MPN-TSS) is a validated tool to objectively measure the burden of symptoms associated with MPN. Baseline TSS will be defined as the average of the daily TSS of 7 consecutive days immediately prior to beginning N-AC. The end of study MPN-TSS will be defined as the average of the daily TSS of 7 consecutive days during week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Fleischman, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California